CLINICAL TRIAL: NCT04592276
Title: The Effects of Lactobacillus Plantarum PS128 on Depression, Anxiety, Cerebral Rhythms, Autonomic Nervous System Function and Sleep Patterns in Self-Reported Insomniacs
Brief Title: The Effects of Lactobacillus Plantarum PS128 in Self-Reported Insomniacs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Yang Ming Chiao Tung University (Other)
Collaborators: Bened Biomedical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: YM107081E
Record Dates: First submitted 2020-10-12; First posted 2020-10-19 (Actual); Last update posted 2022-07-21 (Actual); Status verified 2018-08

CONDITIONS: Insomnia
Keywords: PS128; Anxiety; Depression; Electroencephalography
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Anxiety Disorders; Depression

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PS128 (Experimental): Each PS128 capsule contained 3 × 10^10 colony forming units (CFU) with microcrystalline cellulose and weights 425 ± 25 mg .
  Interventions: Dietary Supplement: PS128
- placebo (Placebo Comparator): The placebo capsules only contained 425 ± 25 mg microcrystalline cellulose.
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: PS128 — Participants took two capsules with PS128 after dinner for 30 days.
  Other Names: Lactobacillus plantarum
  Arms: PS128
Dietary Supplement: placebo — Participants took two capsules without PS128 after dinner for 30 days.
  Arms: placebo

SUMMARY:
To determine whether PS128 (1) reduces the severity of anxiety and depressive symptoms, (2) adjusts autonomic nervous system functioning, and (3) improves sleep quality.

DETAILED DESCRIPTION:
Forty participants with self-reported insomnia between 20 and 40 years old were randomly assigned to two groups, the PS128 and a placebo group, under the double-blind trial. Participants took two capsules with or without PS128 after dinner for 30 days. Study measures included subjective depressive symptoms, anxiety and sleep questionnaires, and miniature polysomnography (miniature-PSG) recordings at baseline and on the 15th and 30th days after taking capsules.

ELIGIBILITY:
Inclusion Criteria:

* (1) aged 20-40 years old,
* (2) 18.5 < BMI < 25,
* (3) BP < 140 mmHg/90 mmHg,
* (4) PSQI >5, ISI>13,
* (5) meet the DSM-5 criteria for chronic primary insomnia.

Exclusion Criteria:

* (1) used other probiotic products within the last two weeks,
* (2) antibiotic treatment within the last month,
* (3) taken sleep medication within the last two months or were on long-term use,
* (4) reported tobacco, alcohol, caffeine or drug addiction,
* (5) lactic acid bacteria allergy,
* (6) cancer, cardiovascular disease, psychiatric illness, kidney disease, diabetes mellitus or other sleep disorders,
* (7) inflammatory bowel disease,
* (8) hepatobiliary gastrointestinal tract surgery
* (9) worked the night shift.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2018-10-11 (Actual); Primary Completion 2019-12-27 (Actual); Study Completion 2019-12-27 (Actual)

PRIMARY OUTCOMES:
Differences in sleep EEG before and after the consumption of probiotics compared to the placebo group. | Baseline, day15 and day30
  According to sleep EEG,we can analysis participants' brain waves (alpha,beta,theta,delta) and sleep stages,etc. to evaluate their objective sleep quality.

SECONDARY OUTCOMES:
Differences in The Beck Depression Inventory II (BDI-II) before and after the consumption of probiotics compared to the placebo group. | Baseline, day15 and day30
  The Beck Depression Inventory II (BDI-II) is a 21-item, self-rated scale that evaluates key symptoms of depression. It rated on a 4-point scale ranging from 0 to 3 based on severity of each item. The maximum total score is 63. A higher score reflects greater symptoms of depression.
Differences in the Beck Anxiety Inventory (BAI) before and after the consumption of probiotics compared to the placebo group. | Baseline, day15 and day30
  the Beck Anxiety Inventory (BAI) is a 21-item, self-rated scale that evaluates anxiety levels , rated on a scale from 0 to 3. Each item is descriptive of subjective, somatic, or panic-related symptoms of anxiety.The maximum total score is 63.A higher score reflects greater anxiety.
Differences in The Pittsburgh Sleep Quality Index (PSQI) before and after the consumption of probiotics compared to the placebo group. | baseline and day30
  The Pittsburgh Sleep Quality Index (PSQI) is a self-report questionnaire that assesses sleep quality over a 1-month time interval. The measure consists of 19 individual items, creating 7 components that produce one global score, and takes 5-10 minutes to complete.The maximum total score is 21. A higher score reflects more poor sleep quality.
Differences in the Insomnia Severity Index (ISI) before and after the consumption of probiotics compared to the placebo group. | Baseline, day15 and day30
  Designed as a brief screening tool for insomnia, the seven-item questionnaire asks respondents to rate the nature and symptoms of their sleep problems using a Likert-type scale. Responses can range from 0 to 4, where higher scores indicate more acute symptoms of insomnia.The maximum total score is 28.
Differences in the Epworth Sleepiness Scale (ESS) before and after the consumption of probiotics compared to the placebo group. | Baseline, day15 and day30
  The Epworth Sleepiness Scale is widely used in the field of sleep medicine as a subjective measure of sleepiness. The test is a list of eight situations in which you rate your tendency to become sleepy on a scale of 0, no chance of dozing, to 3, high chance of dozing.
Differences in heart rate variability (HRV) before and after the consumption of probiotics compared to the placebo group. | Baseline, day15 and day30
  HRV is measured by the variatrasions in the R-R interval between the successive peaks of the QRS complex in the ECG wave. Based on fast Fourier transform, time-domain (R-R interval) transfer to frequency domain resulting total power (TP, 0.0-0.4), low frequency (LF, 0.04-0.15Hz), high frequency (HF, 0.15-0.4Hz), normalized LF (LF%) and LF/HF ratio are obtained. LF% and HF represent an index of sympathetic activity and parasympathetic activity respectively. LF/HF is indicative of the sympathetic to paympathetic autonomic balance.
Differences in Visual Analogue Scale (VAS) before and after the consumption of probiotics compared to the placebo group. | Baseline, day15 and day30
  Visual Analogue Scale (VAS) consists of a line, 10 cm in length. Individuals point to or mark a spot on the line where they feel indicates their current their emotion, fatigue level and sleep quality. The score of emotion level is from 0cm (very nervous) to 10 cm (very relaxing). The score of fatigue level is from 0 cm (very energetic) to 10 cm (very sleepy). The score of sleep quality is from 0 cm (poor) to 10 cm (sleep well). The maximum total score is 100% (equal 10cm).
Differences in the State and Trait Anxiety Index (STAI) before and after the consumption of probiotics compared to the placebo group. | Baseline, day15 and day30
  The State-Trait Anxiety Inventory (STAI) is a psychological inventory based on a 4-point Likert scale and consists of 40 questions on a self-report basis. The STAI measures two types of anxiety - state anxiety, or anxiety about an event, and trait anxiety, or anxiety level as a personal characteristic. The score of state anxiety is from 0 to 80.The score of trait anxiety is from 0 to 80. Higher values represent a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Cheryl C Yang, doctor, Study Chair — Institute of Brain Science ,National Yang-Ming University, Taipei City, Taiwan
Locations (1):
- Institute of Brain Science National Yang Ming University, Taipei, Taiwan